CLINICAL TRIAL: NCT05429099
Title: Virtual Preplanning of Mandibular Reconstruction (ViPMR): a Phase III Randomized Controlled Clinical Trial
Brief Title: Mandibular Reconstruction Preplanning (ViPMR)
Acronym: ViPMR
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Eitan Prisman, Clinical Associate Professor, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: H20-03314
Record Dates: First submitted 2022-06-10; First posted 2022-06-23 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Oral Cavity Cancer; Oral Cancer
Keywords: Oral Cavity Cancer; Oral Cancer; Mandibular Reconstruction
MeSH Terms: conditions — Mouth Neoplasms

STUDY DESIGN:
Intervention Model Description: Both patient groups will receive the standard presurgical work-up including CT imaging, quality of life questionnaires, and a functional evaluation of bite force and jaw mobility.
  Experimental arm - VSP: The trial research engineer (RE) will coordinate with the site surgeon (SS) to create and 3D-print surgical cutting guides for the mandible, for the fibula or scapula, and a 3D computed reconstruction. This reconstruction model will be used to pre-bend a titanium fixation plate. This plate and the surgical cutting guides will be sterilized prior to use. The SS will apply the mandibular cutting guide to make the resection, remove the resected component and apply the pre-bent plate. Next, either the fibular or scapular cutting guide will be applied to harvest the transplant which is then secured to the plate. The flap is re-vascularized using blood vessels in the neck.
  Control arm - FHS: In FHS, the SS will proceed with surgery as per their routine practice.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Free-Hand Surgery (FHS) (Active Comparator): In FHS, the site surgeon will proceed with the surgery as per their routine practice.
  Interventions: Procedure: Free-Hand Surgery
- Virtual Surgical Planning (VSP) (Experimental): The trial research engineer (RE), located at Vancouver General Hospital (VGH), will segment the CT data to create a 3D model for surgical planning. During the teleconference between site surgeon (SS) and RE, the RE will load the CT data and the segmented 3D model into the virtual planning environment. With the RE navigating the software, which was created in-house at VGH and used in a previous case series, the SS will determine the extent of disease and define the resection planes. After the cutting planes are created, the RE will use the software to create the reconstruction plan with either the patient-specific fibula or scapula. Once the surgeon is satisfied with the plan, the teleconference will end and the RE will create and 3D print the surgical guides for the mandible, for the fibula or scapula, as well as the 3D computed reconstruction.
  Interventions: Procedure: Virtual Surgical Planning (VSP)

INTERVENTIONS:
Procedure: Virtual Surgical Planning (VSP) — The 3D reconstruction model, not requiring sterilization, will be sent directly to the SS. Prior to surgery, the SS will prebend a titanium fixation plate to the reconstruction model. Both the surgical cutting guides and titanium plate will be sterilized prior to use in surgery. If the planned resection cannot proceed (possibly due to tumour growth), the surgical team will note the reason for abandonment and conduct a standard FHS. Intraoperatively, the SS will apply the mandibular cutting guide to make the resection, remove the resected component and apply the pre-bent plate. Next, either the fibular or scapular cutting guide is applied to harvest the transplant which is then secured to the plate. The flap is re-vascularized by joining it to blood vessels in the neck.
  Arms: Virtual Surgical Planning (VSP)
Procedure: Free-Hand Surgery — The SS will adopt their standard procedure for the mandibular resection and reconstruction. This typically involves bending a titanium fixation plate, harvesting of the bony flap, and shaping of the segments all intraoperatively based on the SS's judgement.
  Arms: Free-Hand Surgery (FHS)

SUMMARY:
Virtual Surgical Planning (VSP), where 3D modeling is used to create 3D-printed surgical guides, has been shown to improve outcomes for patients who undergo mandibular reconstruction surgery, usually due to invasion of cancer from the oral cavity to the jaw. This trial will directly compare the outcomes of patients who receive VSP versus patients who receive the current standard of care, which is Free-Hand Surgery (FHS). They will be randomized into either treatment at a 1:1 ratio and bony union rates will be compared between 12-month postoperative CT scans for each treatment group. Secondary objectives include comparing other short and long-term complication rates, reconstruction accuracy, quality of life, and functional outcomes of VSP and FHS. An economic analysis of VSP will also be performed.

ELIGIBILITY:
Inclusion Criteria:

* primary diagnosis requiring mandibulectomy and fibular or scapular free flap reconstructive surgery
* are over the age of 18
* cognitive ability and language skills that allow participation in the trial
* provide informed consent

Exclusion Criteria:

* severe comorbidities including metastatic disease
* do not have a recent (within 30 days) CT scan and are unable/unwilling to receive a head CT scan at the latest 6 days prior to surgery
* prior history of head or neck cancer within last 5 years
* prior history of head or neck radiation treatment at any time
* pregnant of lactating women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 420 (Estimated)
Dates: Start 2022-10-15 (Actual); Primary Completion 2025-10-15 (Estimated); Study Completion 2026-10-15 (Estimated)

PRIMARY OUTCOMES:
Bony Union | Assessed on CT scans 12 months postoperatively
  The primary outcome is nonunion as assessed by two independent radiologists at Vancouver General Hospital, blinded to the intervention, based on the 12-month postoperative CT scan. Each apposition (between native bone-flap or between flap segments) will be assessed as nonunion, partial union, and complete union. Cases where there is disagreement between reviewers will undergo consensus review, any persisting disagreements will be reviewed by a third radiologist and classification will be based on the majority vote.

SECONDARY OUTCOMES:
Difference in Intracondylar Distance | Assessed between preoperative CT (at least 6 days prior to surgery) and postoperative CT (5 days after date of surgery) scans
  Comparison to assess structural reconstruction accuracy of postoperative versus preoperative cephalometrics. This will be calculated as the absolute value of postoperative intracondylar distance minus preoperative intercondylar distance (millimeters).
Difference in Mandibular Angles | Assessed between preoperative CT (at least 6 days prior to surgery) and postoperative CT (5 days after date of surgery) scans
  Comparison to assess structural reconstruction accuracy of postoperative versus preoperative cephalometrics. This will calculated as the absolute value of postoperative mandibular angle minus preoperative mandibular angle (degrees).
University of Washington Quality of Life (UWQoL) | Measure documented at time of baseline clinic visit and at 1, 3, 6, 9 and 12 months post-surgery (6 visits total)
  A questionnaire that measures quality of life which records responses on the 5-point Likert scale; minimum of 1 (strongly disagree) and maximum of 5 (strongly agree).
EQ-5D-5L Survey | Measure documented at time of baseline clinic visit and at 1, 3, 6, 9 and 12 months post-surgery (6 visits total)
  Another questionnaire which measures quality of life. Responses recorded as checkboxes that are ticked if applicable to the participant. Participant health is measured on a scale of 0 (worst health imaginable) to 100 (best health imaginable).
Dysphagia | Measure documented at time of baseline clinic visit and at 1, 3, 6, 9 and 12 months post-surgery (6 visits total)
  Measured through responses to the M.D. Anderson Dysphagia Inventory (MDADI) for assessment of dysphagia. MDADI records responses on the 5-point Likert scale; minimum of 1 (strongly disagree) and maximum of 5 (strongly agree).
Oral Health | Measure documented at time of baseline clinic visit and at 1, 3, 6, 9 and 12 months post-surgery (6 visits total)
  Measured through responses to the General Oral Health Assessment Index (GOHAI). Responses recorded one of 5 choices with a point value assigned to each (1 = always, 2 = often, 3 = sometimes, 4 = seldom, and 5 = never).
Fibula harvest site complications | Measure documented at time of baseline clinic visit and at 1, 3, 6, 9 and 12 months post-surgery (6 visits total)
  Measured through responses to the Lower-Limb Tasks Questionnaire (LLTQ) if patient had fibula harvested for reconstruction. or the Disabilities of the Arm, Shoulder, Hand (DASH) questionnaire if patients had scapula harvested for reconstruction. Intends to measure donor site morbidity by assessing ease of task completion (4 = no difficulty, 3 = mild difficulty, 2 = moderate difficulty, 1 = severe difficulty, 0 = unable), as well as importance of task (4 = very important, 3 = moderately important, 2 = mildly important, 1 = not important).
Scapula harvest site complications | Measure documented at time of baseline clinic visit and at 1, 3, 6, 9 and 12 months post-surgery (6 visits total)
  Measured through responses to the Disabilities of the Arm, Shoulder, Hand (DASH) questionnaire if patients had scapula harvested for reconstruction. Intends to measure donor site morbidity by assessing difficulty during tasks (1 = no difficulty, 2 = mild difficulty, 3 = moderate difficulty, 4 = severe difficulty, 5 = unable).
Economic analysis | Measure documented at time of baseline clinic visit and at 1, 3, 6, 9 and 12 months post-surgery (6 visits total)
  Measured through responses to Health Utilization Questionnaire (HUQ) survey to measure impact to patients economic state as a result of their surgery. Records whether participant has experienced certain situations as no or yes (and asks frequency of these situations). Also asks for associated costs that may
Occlusal force (bite force) | Measure documented at time of baseline clinic visit and at 1, 6, and 12 months post-surgery (4 visits total)
  Measured through Dental PreScale System (DPS-Fujifilm Global) as an assessment of patient bite force.
Dental Implantability | Up to 100 days after the post-operative CT scan.
  Oral surgeon on the trial will assess the feasibility of the creation of dental implants for the patient postoperatively; responses will recorded as either feasible (1) or infeasible (0).
Operative Time | Initial Surgery
  Time from first incision to the end of surgical closure as documented on the nursing record.
Ischaemic Time | Initial Surgery
  Time from cutting off blood supply to operative region to restoring blood supply and flow as documented on the nursing record.
Length of Stay | From date of patient's preoperative hospital admission until the date of hospital discharge postoperatively or date of death from any cause, whichever came first, assessed up to 100 days
  Time from admission into hospital preoperatively to discharge from hospital postoperatively as documented on patient's medical chart or date of death, whichever came first.
Rate of Plate Extrusion | Patients will be monitored for 1 year post-operatively
  Complication with plate where may partially or fully be exposed to external environment.
Rate of Flap Failure | Patients will be monitored for 1 year post-operatively
  Complication with flap where donor bone no longer viable as reconstruction piece and replacement required. May be due to ischemic necrosis, infection, osteoradionecrosis, fracturing, etc.
Rate of Cancer Reoccurrence | Patients will be monitored for 1 year post-operatively
  Complication where cancer that was confirmed to be removed (negative resection margins, subsequent chemoradiotherapy results, etc.) reoccurs in the mandibular region. It does not have to be the same type or continuation of previous cancer; any cancer found within mandibular region postoperatively qualifies.
Adverse Events | Charts and interviews reviewed at time of baseline clinic visit and at 1, 3, 6, 9 and 12 months post-surgery (6 visits total)
  Any additional complication or adverse event not covered by other secondary outcomes will be recorded from patient chart review and through a structured interview with the patients.
Occlusion | Measure documented at time of baseline clinic visit and at 1, 6, and 12 months post-surgery (4 visits total)
  Extent of oral occlusion measured during in-person clinic assessments; can be recorded as normal occlusion, malocclusion Class I, malocclusion Class II, or malocclusion Class III.
Jaw Mobility | Measure documented at time of baseline clinic visit and at 1, 6, and 12 months post-surgery (4 visits total)
  Assessment of jaw freedom of movement will be taken during in-person clinic assessments; recorded as measurement of maximal mouth opening (millimeters) from top lip to bottom lip.

CONTACTS AND LOCATIONS:
Locations (1):
- Vancouver General Hospital, Vancouver, British Columbia, Canada

REFERENCES:
- [Derived] Tran KL, Turkdogan S, Dinur AB, Milner TD, Wang E, Nichols A, MacNeil D, Mendez A, Jervis-Bardy J, De Almeida J, Yao C, Goldstein D, Gilbert R, Eskander A, Higgins K, Enepekides D, Gupta M, Zhang H, Au M, Nguyen S, Fels S, Hodgson A, Brasher P, Mitton C, Sabiq F, Fisher C, Yang D, Wong A, Garnis C, Poh C, Durham JS, Prisman E. A multi-centre, participant-blinded, randomized, 3-year study to compare the efficacy of Virtual Surgical Planning (VSP) to Freehand Surgery (FHS) on bony union and quality of life outcomes for mandibular reconstruction with fibular and scapular free flaps: study protocol for a randomized phase II/III trial. BMC Cancer. 2025 Feb 27;25(1):358. doi: 10.1186/s12885-025-13505-5. PMID 40016641